CLINICAL TRIAL: NCT03802409
Title: The Real Word Study of Albumin-binding Taxol for Lung Cancer Treatment
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Anhui Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: AHAT-105
Record Dates: First submitted 2019-01-10; First posted 2019-01-14 (Actual); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Lung Cancer
Keywords: Albumin-binding taxol
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators conduct the real world study to explore the efficacy and safety of Albumin-binding taxol in lung cancer .

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients .
2. Confirmed by Histopathology or Cytology of Lung Cancer
3. Patients should be voluntary to the trial and provide with signed informed consent
4. The researchers believe patients can benefit from the study.

Exclusion Criteria:

1. Patients with a known history of allergic reactions and/or hypersensitivity attributed to Albumin-binding taxol or its accessories
2. Pregnant or lactating women
3. Patients with Albumin-binding taxol contraindications
4. Patients of doctors considered unsuitable for the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Confirmed by Histopathology or Cytology of Lung cancer
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-01-20 (Estimated); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Progress free survival | 1 year
  Progress free survival is defined as the length of time from random assignment to disease progression or to death resulting from any cause other than the progress.

SECONDARY OUTCOMES:
Overall Survival | 3 year
  overall survival is defined as the length of time from random assignment to death or to last contact.
disease control rate | 1 year
  Investigators will assess treatment response according to Response Evaluation Criteria in Solid Tumors 1.1
Objective tumor response rate | 1 year
  Objective tumor response rate is defined as the percentage of subjects having achieved confirmed Complete Response + Partial Response as best overall response according to radiological assessments

OTHER OUTCOMES:
Quality of life score | 1 year
  Quality of life score is a questionnaire developed to assess the quality of life of cancer patients.
adverse events | 1 year
  adverse events are evaluated according to National Cancer Institute Common Terminology Criteria for Adverse Events v4.0.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Within six months after the trial complete.
Access Criteria: The data will be disclosed within six months after completion of the study.